CLINICAL TRIAL: NCT03604159
Title: Buprenorphine Extended-release in Jail and at Re-entry: Open-label Randomized Controlled Trial vs. Daily Sublingual Buprenorphine-naloxone
Brief Title: XRB vs. SLB in Jail and at Re-entry: Pilot, Proof of Concept
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: New York City Health and Hospitals Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-00823
Record Dates: First submitted 2018-07-05; First posted 2018-07-27 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Opioid Dependence
Keywords: Opioid dependence; Buprenorphine; primary care treatment; extended-release buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Sublocade; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Buprenorphine Extended-Release (Experimental): XRB is a 300mg pre-mixed subcutaneous injectable formulation to be administered monthly. XRB is for abdominal subcutaneous injection only. Participants in the XRB treatment arm will be given 1 or more XRB injections prior to release from jail and one more at week 5 post-release, depending on their release date.
  Interventions: Drug: Buprenorphine Extended Release
- Sublingual Buprenorphine (Active Comparator): SLB (SUBOXONE, Zubsolv, or generic tablets) is a daily sublingual film or tablet ranging from 8-24mg/day or equivalent (Zubsolv is dosed 5.7-17.1 mg/day). The film or tablet is placed under the tongue for 5 to 10 minutes until dissolved completely. Participants in the SLB treatment arm will be provided SLB daily by observed dosing in-jail (controlled substances are not self-administered in-jail) and and encouraged to continue SLB treatment in weekly, bi-weekly, or monthly quantities for unobserved, daily, self-administration through week 5. Patients may also elect to obtain SLB care free-of-charge from the Bellevue Hospital Center Addiction Medicine clinic or from non-NYU/Bellevue providers and pharmacies per usual care standards. SLB will not be provided via the study.
  Interventions: Drug: Sublingual Buprenorphine (SUBOXONE, Zubsolv, or generic tablets)

INTERVENTIONS:
Drug: Buprenorphine Extended Release — XRB is available in dosage strengths of 100 mg/0.5 mL and 300 mg/1.5 mL buprenorphine. Each dose is provided in a prefilled syringe with a 19 gauge 5/8-inch needle.
  Other Names: SUBLOCADE
  Arms: Buprenorphine Extended-Release
Drug: Sublingual Buprenorphine (SUBOXONE, Zubsolv, or generic tablets) — SLB is administered sublingually or buccally as a single daily dose. Medication should be prescribed in consideration of the frequency of visits. Provision of multiple refills is not advised in early treatment or without appropriate follow-up visits. After treatment induction and stabilization, the maintenance dose of SLB is generally in the range of 4mg/1mg buprenorphine/naloxone to 24mg/6mg buprenorphine/naloxone per day depending on the individual patient and clinical response.
  Arms: Sublingual Buprenorphine

SUMMARY:
This is a pilot proof-of-concept randomized controlled trial, open-label and unblinded, examining the feasibility and acceptability of Buprenorphine extended-release vs. daily sublingual buprenorphine-naloxone for the treatment of opioid use disorder in jail and at community re-entry.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18yo incarcerated in NYC jails with known release dates.
* DSM-V criteria for current opioid use disorder (DSM-IV opioid dependence).
* Currently maintained on sublingual buprenorphine-naloxone in the NYC jail opioid treatment program.

Exclusion Criteria:

* Individual not interested in XRB treatment. Current SLB patients are otherwise by definition appropriate for XRB.
* Pregnant or planning conception. A urine dipstick pregnancy (hCG) test will be administered at baseline. The test detects human chorionic gonadotropin (hCG) in urine with a sensitivity/specificity of: 25 mIU hCG/ml, >99%. Time to result is four minutes. If negative, a urine pregnancy test will be administered bi-weekly thereafter to ensure that a participant is not pregnant
* No severe or acute medical or psychiatric disability preventing safe study participation or making follow-up unlikely.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Lee, MD, MSc, Principal Investigator — NYU School of Medicine
Locations (1):
- Bellevue Hospital Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting requests and accessing data may be found at (Link to be provided).
Supporting Information: Study Protocol, ICF
Time Frame: To achieve aims in the approved proposal.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Cheng A, Badolato R, Segoshi A, McDonald R, Malone M, Vasudevan K, Badiei B, Sugarman A, Macdonald R, Mangat J, Giftos J, Lee JD, Tofighi B. Perceptions and experiences toward extended-release buprenorphine among persons leaving jail with opioid use disorders before and during COVID-19: an in-depth qualitative study. Addict Sci Clin Pract. 2022 Jan 29;17(1):4. doi: 10.1186/s13722-022-00288-4. PMID 35093164
- [Derived] Lee JD, Malone M, McDonald R, Cheng A, Vasudevan K, Tofighi B, Garment A, Porter B, Goldfeld KS, Matteo M, Mangat J, Katyal M, Giftos J, MacDonald R. Comparison of Treatment Retention of Adults With Opioid Addiction Managed With Extended-Release Buprenorphine vs Daily Sublingual Buprenorphine-Naloxone at Time of Release From Jail. JAMA Netw Open. 2021 Sep 1;4(9):e2123032. doi: 10.1001/jamanetworkopen.2021.23032. PMID 34495340

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Buprenorphine Extended-Release | Sublingual Buprenorphine
Started | 26 | 26
Completed | 20 | 19
Not Completed | 6 | 7
Not completed — Lost to Follow-up | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine Extended-Release | Sublingual Buprenorphine | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (9.2) | 42.3 (10.8) | 42.7 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 23 | 22 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 9 | 23
  Not Hispanic or Latino | 12 | 17 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 9 | 15
  White | 7 | 12 | 19
  More than one race | 13 | 4 | 17
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: # of Participants Retained on Any Form of Community Buprenorphine (Not Randomzied tx) at Week 8
Description: Retained on any form of community buprenorphine treatment at Week 8
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine Extended-Release | Sublingual Buprenorphine
Number analyzed (Participants) | 26 | 26
Participants | 18 | 9

2. Primary Outcome: # of Participants Retained on Their Randomly Assigned Treatment at Week 8
Description: Retained on assigned treatment at Week 8
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine Extended-Release | Sublingual Buprenorphine
Number analyzed (Participants) | 26 | 26
Participants | 15 | 9

3. Primary Outcome: Mean # of Weeks (0-8) on Any Buprenorphine Treatment
Description: Weeks (0-8) on buprenorphine treatment, mean (SD)
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Buprenorphine Extended-Release | Sublingual Buprenorphine
Number analyzed (Participants) | 26 | 26
weeks | 6.1 (3.5) | 2.6 (3.2)

4. Primary Outcome: Urine Samples Opioid-negative
Description: number of opioid-negative urine samples
Time Frame: 8 weeks
Measure: Number; unit: urine samples
Units Other Than Participants: Urine Tests
Arm/Group | Buprenorphine Extended-Release | Sublingual Buprenorphine
Number analyzed (Participants) | 26 | 26
Number analyzed (Urine Tests) | 100 | 100
urine samples | 72 | 50

5. Primary Outcome: the # of Participants Re-incarcerated
Description: Re-incarceration
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine Extended-Release | Sublingual Buprenorphine
Number analyzed (Participants) | 26 | 26
Participants | 2 | 4

6. Primary Outcome: The Mean In-jail Medical Visits Per Day Following Randomization and Induction on Study Medication
Description: Jail medical clinic visits per day following study medication induciton, mean
Time Frame: Post-randomization and pre-release, (0-3 months)
Measure: Mean (Full Range); unit: jail clinic visits per day
Arm/Group | Buprenorphine Extended-Release | Sublingual Buprenorphine
Number analyzed (Participants) | 26 | 26
jail clinic visits per day | 0.11 [.05 to 0.16] | 1.06 [0.88 to 1.23]

7. Secondary Outcome: The # of Participants That Received Their Randomly Assigned Study Medication
Description: Received assigned study medication
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine Extended-Release | Sublingual Buprenorphine
Number analyzed (Participants) | 26 | 26
Participants | 24 | 26

8. Secondary Outcome: The # of Participants Who Received Their Randomly Assigned Study Medication Prior to Release From Jail as Scheduled
Description: Received assigned study medication prior to release as scheduled
Time Frame: 0-3 months (pre-release)
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine Extended-Release | Sublingual Buprenorphine
Number analyzed (Participants) | 26 | 26
Participants | 21 | 26

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Buprenorphine Extended-Release | Sublingual Buprenorphine
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 2/26 | 0/26
Other Adverse Events (participants affected / at risk) | 5/26 | 3/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine Extended-Release (N=26) | Sublingual Buprenorphine (N=26)
Foot Infection (Infections and infestations) | 1 (1) | 0 (0)
Toe Amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine Extended-Release (N=26) | Sublingual Buprenorphine (N=26)
Stomach flu (General disorders) | 0 (0) | 1 (1)
Kidney Stones (Renal and urinary disorders) | 1 (1) | 0 (0)
Nausea/Fatigue (General disorders) | 1 (1) | 0 (0)
intoxication induction (General disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Sinus infection (Infections and infestations) | 0 (0) | 1 (1)
soreness at injection site (General disorders) | 1 (1) | 0 (0)
Pain in upper-left arm (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT03604159/Prot_SAP_000.pdf